CLINICAL TRIAL: NCT04742998
Title: Validity of a Task of Acoustic-phonetic Decoding on Anatomic Deficits in Paramedical Assessment of Speech Disorders for Patients Treated for Oral or Oropharyngeal Cancer
Brief Title: Task of Acoustic-phonetic Decoding on Anatomic Deficits in Paramedical Assessment of Speech Disorders for Patients Treated for Oral or Oropharyngeal Cancer
Acronym: DAPADAF-E
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Laboratoire parole et langage (Unknown); Laboratoire Information Avignon université (Unknown); IRIT - Institut de Recherche en Informatique de Toulouse (Unknown)
Responsible Party: Sponsor
Other Study IDs: RC31/20/0551; 2020-A02335-34 (Other: ID-RCB)
Record Dates: First submitted 2021-02-02; First posted 2021-02-08 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Speech Intelligibility
Keywords: speech deficit; tumor pathologies of the upper aero-digestive tract
MeSH Terms: conditions — Speech Intelligibility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated for an oral or oropharyngeal tumor for at least 6 months: Patients treated for an oral or oropharyngeal tumor for at least 6 months
  Interventions: Other: Acoustic-phonetic decoding task (DAP)

INTERVENTIONS:
Other: Acoustic-phonetic decoding task (DAP) — Completion of speech-related quality of life autoquestionnaires Routine speech assessment Acoustic-phonetic decoding task (DAP) two lists of 16 pseudo-words

SUMMARY:
The bridging of the gap between speech production and perception by the interlocutor would be made possible by the use of a more suitable and automatic task. An acoustic-phonetic decoding test (or DAP in French, i.e. the production of isolated pseudo-words in repetition or reading), created within the framework of the The French National Cancer Institute (InCA) C2SI project, avoids the effects of cognitive restoration by the interlocutor. An automatic score from the DAP would lead to an overall score per patient, but also to scores specific to each phonetic segment, to be correlated with the analytical scores from each anatomical oropharyngeal segment.

The study hypothesis is that the automatic processing of an acoustic-phonetic decoding task during the assessment in current practice is a valid and reliable tool for diagnosing oropharyngeal analytical and dynamic deficits by highlighting deficient linguistic units.

The study hypothesis is that the automatic processing of an acoustico-phonetic decoding task during the assessment in current practice is a tool for diagnosing oropharyngeal analytical and dynamic deficits by highlighting deficient linguistic units.

DETAILED DESCRIPTION:
Fifth cancer in terms of incidence in France, tumor pathologies of the upper aero-digestive tract, due to their location, impact the speech abilities of affected subjects. Speech therapy in paramedical clinical assessments consist of two parts.

* The analytical part to highlight the anatomical and dynamic deficits of segments involved in speech.
* The functional part characterizes the pathophysiological impact by means of an "ear" assessment.

The link between anatomy and functional speech deficit is very close in oncology (the location and the size of the tumor, the structural changes due to the treatment who modify the oropharyngeal dynamics and the mechanisms involved in the production of the speech), but the correlation is weak between functional intelligibility scores and analytical motor scores. Indeed, the perception of speech by a human listener is not a simple "recording" of the production, but a representation of this production after implementation of individual mechanisms for restoring the acoustic information linked to the lexicon or to the context by the listener. The listener's degree of familiarity with the speaker or his pathology is also a source of variability.

The bridging of the gap between speech production and perception by the interlocutor would be made possible by the use of a more suitable and automatic task. An acoustic-phonetic decoding test (or DAP in French, i.e. the production of isolated pseudo-words in repetition or reading), created within the framework of the InCA C2SI project, avoids the effects of cognitive restoration by the interlocutor. An automatic score from the DAP would lead to an overall score per patient, but also to scores specific to each phonetic segment, to be correlated with the analytical scores from each anatomical oropharyngeal segment.

The study hypothesis is that the automatic processing of an acoustic-phonetic decoding task during the assessment in current practice is a valid and reliable tool for diagnosing oropharyngeal analytical and dynamic deficits by highlighting deficient linguistic units.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged at least 18 years old and benefiting from a social security scheme
* Native French-speaking patients
* Patients treated for cancer of the oral cavity or oropharynx (surgical and / or radiotherapy and / or chemotherapy treatment)
* Patients in clinical remission for at least 6 months (chronic nature and stability of the disorders)
* All tumor sizes according to the tumor (T), node (N), and metastasis (M) categories (TNM classification) (T1 to T4)
* Patients with a perceptible speech disorder in a conversational situation or not (to allow the determination of fine deficits)
* Patients who do not object to carrying out the research

Exclusion Criteria:

* Patients with an associated pathology potentially responsible for speech or fluency disorders (joint, speech and language disorders of developmental, organic or functional origin, voice disorders of organic or functional origin, stammering , stammering, fluency disturbances, speech disturbances of neurological origin)
* Patients reporting an auditory complaint and not having a hearing aid
* Inability to provide the person with enlightened information and to ensure the subject's compliance because of impaired physical and / or psychological health,
* Patients participating in another research including an exclusion period still in progress.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All site have an active group of person allowing a feasibility of recruitment
Sampling Method: Non-Probability Sample
Enrollment: 116 (Estimated)
Dates: Start 2021-10-22 (Actual); Primary Completion 2024-10-22 (Estimated); Study Completion 2024-10-22 (Estimated)

PRIMARY OUTCOMES:
Correlation coefficient | Day 1
  Correlation coefficient between he automatic score by phoneme class from the DAP and the score for each oropharyngeal anatomical segment from muscle testing

SECONDARY OUTCOMES:
Human perceptual score - Direct transcription | Day 1
  the speech therapist will transcribe the pseudo-word he thinks he has recognized immediately after the subject says it, using software installed on the examination computer. A perceptual score of linguistic traits of average difference (between expected production and perception by the speech therapist) by phoneme will then be determined.
Human perceptual score - jury transcription | Day 1
  Audio recordings of the task will be made. A perceptual score of linguistic traits of average difference (between expected production and perception by the jury) by phoneme will then be determined
Head and Neck Carcinologic Handicap Index (HNCHI) | Day 1
  Correlation between HNCHI and scores from the DAP

CONTACTS AND LOCATIONS:
Overall Officials: Clémence DEVOUCOUX, Principal Investigator — University Hospital, Toulouse
Locations (3):
- France (3):
  - AP- H Marseille - Hôpital de la Conception, Marseille
  - Institut universitaire du Cancer de Toulouse - Oncopole, Toulouse
  - University Hospital Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balaguer M, Farinas J, Fichaux-Bourin P, Puech M, Pinquier J, Woisard V. Validation of the French Versions of the Speech Handicap Index and the Phonation Handicap Index in Patients Treated for Cancer of the Oral Cavity or Oropharynx. Folia Phoniatr Logop. 2020;72(6):464-477. doi: 10.1159/000503448. Epub 2019 Nov 15. PMID 31734664
- [Background] Balaguer M, Champenois M, Farinas J, Pinquier J, Woisard V. The (head and neck) carcinologic handicap index: validation of a modular type questionnaire and its ability to prioritise patients' needs. Eur Arch Otorhinolaryngol. 2021 Apr;278(4):1159-1169. doi: 10.1007/s00405-020-06201-6. Epub 2020 Jul 14. PMID 32666294
- [Background] Lalain M, Ghio A, Giusti L, Robert D, Fredouille C, Woisard V. Design and Development of a Speech Intelligibility Test Based on Pseudowords in French: Why and How? J Speech Lang Hear Res. 2020 Jul 20;63(7):2070-2083. doi: 10.1044/2020_JSLHR-19-00088. Epub 2020 Jun 29. PMID 32598209